CLINICAL TRIAL: NCT05505565
Title: Continuous Glucose Monitors in the Management of Youth With Prediabetes
Brief Title: Tolerability, Acceptance, and Utility of Intermittent CGM Use in Youth With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jessica Schmitt, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009480; P30DK079626 (NIH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: PreDiabetes; Obesity; Insulin Resistance
Keywords: pediatrics; prediabetes; obesity
MeSH Terms: conditions — Prediabetic State; Obesity; Insulin Resistance | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized, non-blinded, parallel, intervention vs control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CGM + Traditional Counseling (Experimental): Subjects in this arm will receive intermittent CGM to be used for 2-weeks each month for the 6-month study period. They will be required to wear a CGM during baseline, 3-month, and 6-month periods. Additional CGM sensors will be supplied for months 1, 2, 4, and 5 and will be optional. They will be provided with a Sworkit(R) account to monitor physical activity completed through the Sworkit(R) website/platform.
  Interventions: Device: Abbott Freestyle Libre 2; Other: Standard physical activity and nutritional counseling for prediabetes management
- Control (Active Comparator): Subjects in this arm will receive standard medical care for pre-diabetes. They will be provided with a Sworkit(R) account to monitor physical activity completed through the Sworkit(R) website/platform.
  Interventions: Other: Standard physical activity and nutritional counseling for prediabetes management

INTERVENTIONS:
Device: Abbott Freestyle Libre 2 — Subjects will be educated on use of Abbott Freestyle Libre 2 and educated on how daily activities impact glucose.
  Arms: CGM + Traditional Counseling
Other: Standard physical activity and nutritional counseling for prediabetes management — Subjects will be advised on recommendations for nutrition and activity goals for preventing progression of prediabetes.

SUMMARY:
We are evaluating whether intermittent use of continuous glucose monitors (CGMs) in addition to standard nutritional counseling and physical activity counseling is associated with improved metabolic health for youth with pre-diabetes (PD).

DETAILED DESCRIPTION:
The purpose of this research study is to test if CGMs are tolerable to youth with pre-diabetes (PD) and their caregivers. We are also evaluating if CGMs add benefit to standard treatment in youth with prediabetes. The CGM in question, Abbott Freestyle Libre 2 is approved by the Food and Drug Administration (FDA) to treat patients aged 4 and up with diabetes. We want to determine if this CGM may benefit people who have PD. People who enter the study will either receive standard medical care for prediabetes or receive standard medical care for prediabetes plus use a CGM for 2 weeks each month to receive real-time biofeedback on their glucose levels during the day.

There will be 3 visits over a 6-month period, baseline, 3-month, and 6-month visits. At each visit fasting labs will be obtained including: complete metabolic panel, lipid panel, pro-insulin, c-peptide, insulin. Anthropomorphics including body mass index, waist circumference, and hip circumference will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age 11 or older
* English-speaking
* stable metformin dose for 1 month prior to enrollment or no metformin use
* baseline A1c of 5.7-6.4%
* BMI > = 85% for age

Exclusion Criteria:

* BMI < 85% for age
* chronic steroid use
* diagnosis of type 1 diabetes, type 2 diabetes, other forms of diabetes
* current or history of malignancy

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
CGM Acceptability | 6 months
  Caregiver and patient acceptability of CGM use
Progression of prediabetes | 6 months
  change in hemoglobin A1c

SECONDARY OUTCOMES:
Insulin sensitivity | 6 months
  HOMA-IR, fasting c-peptide, fasting pro-insulin
Hyperlipidemia | 6 months
  LDL, triglyceride, HDL, total cholesterol measurements
Transaminitis | 6 months
  AST, ALT
Glycemic metrics | 6 months
  CGM data including: time in target range, time above target range, post-prandial glucose excursion

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Schmitt, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No